CLINICAL TRIAL: NCT07156344
Title: An Observational Cohort Study on the Identification and Outcome Evaluation of Intracranial Atherosclerotic Plaque Vulnerability
Brief Title: Assessing Vulnerability and Outcomes of Intracranial Atherosclerotic Plaques
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The People's Hospital of Liaoning Province (Other); The First Hospital of Jilin University (Other); Jilin Electric Power Hospital (Unknown); Jilin city central hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-417-002
Record Dates: First submitted 2025-06-11; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Asymptomatic Intracranial Atherosclerotic Stenosis Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic Intracranial Atherosclerotic Patients
  Interventions: Diagnostic Test: Progression and Outcome of Intracranial Atherosclerosis

INTERVENTIONS:
Diagnostic Test: Progression and Outcome of Intracranial Atherosclerosis — "Progression and Outcome of Intracranial Atherosclerosis" is the primary endpoint; all others are secondary endpoints. Stroke defined as any stroke and new ipsilateral stroke (including ischemic and hemorrhagic stroke) associated with vascular stenosis.
  Other Names: Medically confirmed death; Myocardial infarction; Onset and Progression of Cognitive Impairment; Worsening of functional outcomes (mRS score ≥2); Stroke was identified on imaging

SUMMARY:
This prospective cohort study aims to establish a large-scale cohort for primary stroke prevention in asymptomatic intracranial atherosclerosis (ICAS). Objectives include: characterizing risk factor and stenotic artery distributions; determining optimal TCD screening sentinel arteries; observing plaque progression/regression via HR-MRI; establishing vulnerable plaque evaluation systems through stroke event follow-up; and developing cognitive decline prediction models integrating hemodynamic parameters. All procedures (TCD, HR-MRI, neuropsychological assessments) are routine clinical examinations with minimal risk. Participation is voluntary. Initial TCD and qualifying HR-MRI scans incur standard fees; all follow-up imaging and neuropsychological assessments post-enrollment are provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial arterial stenosis confirmed by transcranial Doppler (TCD), clinically suspected to be of atherosclerotic origin
* No history of stroke or transient ischemic attack (TIA)
* Adequate temporal bone acoustic window penetrability

Exclusion Criteria:

* Clinically diagnosed non-atherosclerotic etiology-related intracranial arterial stenosis
* Poor temporal bone acoustic window penetrability
* Loss to follow-up

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Transcranial Doppler (TCD)-detected asymptomatic intracranial atherosclerotic patients
Sampling Method: Non-Probability Sample
Enrollment: 3849 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with Progression of Intracranial Atherosclerosis | 4 years
  Number of participants with Progression of intracranial atherosclerosis encompass intracranial arterial stenosis, development of new stenoses, worsening of existing stenoses, as well as decrease, regression, or resolution of stenosis.

SECONDARY OUTCOMES:
Number of participants with Clinical adverse event | 4 years
  Clinical adverse events include stroke, death, myocardial infarction, onset and progression of cognitive impairment and worsening of functional outcomes (mRS score ≥2)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen HX, Wang LJ, Yang Y, Yue FX, Chen LM, Xing YQ. The prevalence of intracranial stenosis in patients at low and moderate risk of stroke. Ther Adv Neurol Disord. 2019 Aug 13;12:1756286419869532. doi: 10.1177/1756286419869532. eCollection 2019. PMID 31447935
- [Background] Wang YJ, Li ZX, Gu HQ, Zhai Y, Zhou Q, Jiang Y, Zhao XQ, Wang YL, Yang X, Wang CJ, Meng X, Li H, Liu LP, Jing J, Wu J, Xu AD, Dong Q, Wang D, Wang WZ, Ma XD, Zhao JZ; China Stroke Statistics Writing Committee. China Stroke Statistics: an update on the 2019 report from the National Center for Healthcare Quality Management in Neurological Diseases, China National Clinical Research Center for Neurological Diseases, the Chinese Stroke Association, National Center for Chronic and Non-communicable Disease Control and Prevention, Chinese Center for Disease Control and Prevention and Institute for Global Neuroscience and Stroke Collaborations. Stroke Vasc Neurol. 2022 Oct;7(5):415-450. doi: 10.1136/svn-2021-001374. Epub 2022 Apr 20. PMID 35443985
- [Background] GBD 2021 Stroke Risk Factor Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Neurol. 2024 Oct;23(10):973-1003. doi: 10.1016/S1474-4422(24)00369-7. PMID 39304265